CLINICAL TRIAL: NCT04933344
Title: Pharmacokinetics and Toxicodynamics of Daptomycin in Bone and Joint Infections
Acronym: PKTOXDAP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Hospices Civils de Lyon (Other)
Responsible Party: Sponsor
Other Study IDs: 397
Record Dates: First submitted 2021-06-15; First posted 2021-06-21 (Actual); Last update posted 2022-05-06 (Actual); Status verified 2022-05

CONDITIONS: Dactinomycin Adverse Reaction; Bone and Joint Infection
Keywords: bone and joint infection; adverse event; daptomycin; Eosinophilic pneumonia; CPK; rhabdomyolysis
MeSH Terms: conditions — Pulmonary Eosinophilia; Rhabdomyolysis | interventions — Daptomycin

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- patients having had BJI or PJI treated with daptomycin: patients having an osteoarticular infection treated with daptomycin and which developped eosinophilic pneumonia or elevation of CPK
  Interventions: Other: patients having had BJI or PJI treated with daptomycin

INTERVENTIONS:
Other: patients having had BJI or PJI treated with daptomycin — patients having had BJI or PJI treated with daptomycin who developped an adverse event : eosinophilic pneumonia and/or elevation of CPK

SUMMARY:
the aim of this study is to investigate the relationship between exposure to daptomycin and the occurrence of muscle toxicity or eosinophilic pneumonia in patients treated with daptomycin for bone and joint infection

DETAILED DESCRIPTION:
Daptomycin is widely used in osteoarticular infections (IOA), as an alternative to vancomycin, and recommended for this use by various learned societies including the Infectious Diseases Society of America (IDSA) in 2013.

Tolerance to daptomycin is generally favorable, with in particular better renal tolerance than vancomycin. However, two rare and potentially severe side effects have been described with this antibiotics: muscle toxicity and eosinophilic pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have had an osteoarticular infection, treated with daptomycin, with at least one blood test for daptomycin performed

Exclusion Criteria:

* Patients who objected to participating in the study
* Absence of blood dosage of daptomycin

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients managed at the CRIOAc Lyon who have had an osteoarticular infection, treated with daptomycin, with at least one blood test for daptomycin performed
Sampling Method: Non-Probability Sample
Enrollment: 1130 (Estimated)
Dates: Start 2021-06-15 (Actual); Primary Completion 2022-03-01 (Actual); Study Completion 2022-07-01 (Estimated)

PRIMARY OUTCOMES:
rate of patients having had a PJI or BJI treated by daptomycin | between 2010 and 2020
  proportion of patients treated by daptomycin
description of BJI/PJI | between 2010 and 2020
  type of BJI or PJI
description of patients | between 2010 and 2020
  comorbidites
description of adverse event | between 2010 and 2020
  type of adverse event
rate of patients having had an adverse event | between 2010 and 2020
  proportion of patients having had an adverse event under daptomycin
Evalutation of the adverse event due to daptomycin : dosage of daptomycine | between 2010 and 2020
  description of the use of daptomycine : dosage
Evalutation of the adverse event due to daptomycin : duration of daptomycine | between 2010 and 2020
  description of the use of daptomycine : duration
Evalutation of the adverse event due to daptomycin : daptomycine plasma clearance | between 2010 and 2020
  mean daptomycine plasma clearance (unit, liters per hour)
Evalutation of the adverse event due to daptomycin : daptomycine volume distribution | between 2010 and 2020
  mean daptomycine volume of distribution (unit, liters)

CONTACTS AND LOCATIONS:
Locations (1):
- Hospices Civils de Lyon, Lyon, France

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://www.crioac-lyon.fr/